CLINICAL TRIAL: NCT01166243
Title: A Phase III Randomized, Controlled, Superiority Study Evaluating the Fibrin Pad Versus Standard of Care Treatment in Controlling Parenchymal Bleeding During Elective Hepatic Surgery
Brief Title: The Fibrin Pad Liver Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Collaborators: OMRIX Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 400-10-001; 2010-019427-58 (EudraCT Number)
Record Dates: First submitted 2010-07-06; First posted 2010-07-21 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Hemorrhage
Keywords: Hemostasis
MeSH Terms: conditions — Hemorrhage | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fibrin Pad (Experimental): Biologic
  Interventions: Biological: Fibrin Pad
- Standard of Care (Other): Procedure
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Biological: Fibrin Pad — Fibrin Pad is a sterile bio-absorbable combination product consisting of two constituent parts- a flexible matrix and a coating of two biological components (Human Fibrinogen and Human Thrombin).
  Arms: Fibrin Pad
Procedure: Standard of Care — Standard of Care is a composite of techniques/methods typically used by the surgeon to control bleeding.
  Arms: Standard of Care

SUMMARY:
The objective of this study is to evaluate the safety and and hemostatic effectiveness of the Fibrin Pad (FP) versus standard of care treatment (SoC) in controlling parenchymal bleeding during hepatic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects > 18 years of age, requiring elective or urgent, open hepatic surgery
* Presence of an appropriate bleeding hepatic parenchymal Target Bleeding Site (TBS) as identified intra-operatively by the surgeon
* Subjects must be willing to participate in the study, and provide written informed consent

Exclusion Criteria:

* Subjects with any intra-operative findings identified by the surgeon that may preclude conduct of the study procedure
* TBS is from large defects in arteries or veins where the injured vascular wall requires repair with maintenance of vessel patency and which would result in persistent exposure of the FP to blood flow and pressure during healing and absorption of the product
* TBS with major arterial bleeding requiring suture or mechanical ligation
* Subjects admitted for trauma surgery
* Subject is a transplant patient for fulminant hepatic failure
* Subject with TBS within an actively infected field
* Bleeding site is in, around, or in proximity to foramina in bone, or areas of bony confine
* Subjects with known intolerance to blood products or to one of the components of the study product or is unwilling to receive blood products
* Subjects who are known, current alcohol and / or drug abusers
* Subjects who have participated in another investigational drug or device research study within 30 days of surgery
* Female subjects who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2010-07; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving hemostasis at the Target Bleeding Site (TBS). | Intra-operative

SECONDARY OUTCOMES:
Proportion of subjects achieving hemostasis success at 10-minutes following randomization. | Intra-operative
Absolute time to hemostasis | Intraoperative
Subjects requiring re-treatment | Intraoperative
Incidence of adverse events potentially related to re-bleeding at TBS | Intraoperative through 60 days
Incidence of adverse events potentially related to thrombotic events | Intraoperative through 60 days
Incidence of adverse events | Intraoperative through 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Hammond, MD, Study Director — Ethicon, Inc.
Locations (9):
- Australia (3):
  - Flinders Medical Centre, Bedford Park, South Australia
  - Queen Elizabeth Hospital, Woodville, South Australia
  - The Alfred, Melbourne, Victoria
- University Hospital of the University of Saarland, Straße, Germany
- University Medical Center, Groningen, Netherlands
- Auckland City Hospital, Grafton, New Zealand
- United Kingdom (3):
  - Queen Elizabeth Hospital, Birmingham
  - Addenbrookes Hospital, Cambridge
  - Royal Infirmary of Edinburgh, Edinburgh

REFERENCES:
- [Result] Koea JB, Batiller J, Patel B, Shen J, Hammond J, Hart J, Fischer C, Garden OJ. A phase III, randomized, controlled, superiority trial evaluating the fibrin pad versus standard of care in controlling parenchymal bleeding during elective hepatic surgery. HPB (Oxford). 2013 Jan;15(1):61-70. doi: 10.1111/j.1477-2574.2012.00583.x. Epub 2012 Oct 16. PMID 23216780
- [Derived] Corral M, Ferko N, Hollmann S, Hogan A, Jamous N, Batiller J, Shen J. Clinician reported ease of use for a novel fibrin sealant patch for hemostasis: results from four randomized controlled trials. Curr Med Res Opin. 2016;32(2):367-75. doi: 10.1185/03007995.2015.1128405. Epub 2015 Dec 21. PMID 26636489